CLINICAL TRIAL: NCT01867255
Title: Pharmacokinetic Study Comparing Area Under the Curve for a Single Dose of Venlafaxine ER Pre- and Post-gastric Bypass
Brief Title: Study to Examine the Effect of Gastric Bypass Surgery on Venlafaxine ER Blood Levels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Carrie A. Krieger, PharmD, BCACP, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12-005860
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Bariatric Surgery; Gastric Bypass; Roux-en-Y Gastric Bypass
Keywords: venlafaxine; Effexor; antidepressive agent
MeSH Terms: interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- venlafaxine ER (Other): venlafaxine ER (extended-release) 75 mg once
  Interventions: Drug: venlafaxine ER (extended-release) 75 mg

INTERVENTIONS:
Drug: venlafaxine ER (extended-release) 75 mg — A single dose of venlafaxine ER 75 mg is to be administered once at each of two study visits, pre- and post-gastric bypass surgery.
  Other Names: Effexor XR 75 mg

SUMMARY:
The purpose of the study is to determine whether a significant and predictable change in bioavailability of extended-release venlafaxine occurs following Roux-en-Y gastric bypass.

ELIGIBILITY:
Inclusion criteria:

- Approved to undergo Roux-en-Y gastric bypass surgery (cost of surgery is NOT included in the study)

Exclusion criteria:

* Pregnant
* Allergy to venlafaxine or desvenlafaxine
* Psychiatric hospitalization within the prior 12 months
* Active professional treatment for recent substance abuse within 12 months of abstinence
* Ongoing psychologic issues, such as personality disorders, difficulties as a trauma survivor, or difficulties with depression unless a stable, documented course of treatment by a licensed mental health professional is available
* Current use of any of the following medications/supplements: 5-hydroxytryptophan, almotriptan, amitriptyline, amoxapine, amoxicillin-clavulanate, amphetamine-dextroamphetamine, atazanavir, bupropion, cinacalcet, citalopram, clarithromycin, clomipramine, desipramine, desvenlafaxine, dextroamphetamine, dextromethorphan, doxepin, duloxetine, eletriptan, entacapone, escitalopram, fluoxetine, fluvoxamine, frovatriptan, haloperidol, imipramine, isocarboxazid, itraconazole, jujube seed extract, linezolid, maprotiline, methylene blue, metoclopramide, metoprolol, milnacipran, mirtazapine, naratriptan, nefazodone, nelfinavir, nortriptyline, paroxetine, phenelzine, procarbazine, protriptyline, quinidine, rasagiline, ritonavir, rizatriptan, saquinavir, selegiline, sertraline, St. John's wort, sumatriptan, tapentadol, terbinafine, toremifene, tramadol, tranylcypromine, trazodone, trifluoperazine, trimipramine, tryptophan, L-tryptophan, venlafaxine, vilazodone, zolmitriptan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Venlafaxine levels pre- and post-gastric bypass | 3 to 4 months
  This study will measure and compare venlafaxine and desvenlafaxine levels in participants before, and again 3 to 4 months after, gastric bypass surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Krieger, PharmD, RPh, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States